CLINICAL TRIAL: NCT03142711
Title: Validation of a Mobile Phone Based on EPRO Tool in Subjects With Systemic Lupus Erythematosus
Acronym: VALUE
Status: Completed | Type: Observational
Sponsor: Lupus Research Alliance (Other)
Collaborators: Pfizer (Industry); Ampel BioSolutions, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AMP-003
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: SLE; Lupus Erythematosus, Systemic; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Medical Intervention — Validation of phone ePRO

SUMMARY:
Systemic lupus erythematosus (SLE) may involve a variety of organ systems expressed differently from patient to patient, and so can be difficult to characterize clinically. Patient reported outcomes (PROs), which consist of feedback directly from patients regarding their symptoms without interpretation by a clinician, are typically used in SLE to supplement other clinical measures. Standard PROs typically used in SLE include the 36-item short form health survey (SF-36), the functional assessment of chronic illness therapy - fatigue (FACIT-F), and the patient global assessment (PtGA), administered by paper or electronic tablet during the clinic visits. The recent development of electronic mobile device technology, such as the smartphone, has made it possible to collect PRO information away from the clinical site in the subject's environment. This study will assess by measurement equivalence testing whether data collected via a smartphone are comparable to that collected in standard fashion and whether PROs obtained in the subject's environment may be more informative than that collected in the physician's office on paper.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Males or females, aged 18 years or older
3. Classification of SLE by either the American College of Rheumatology (ACR) or Systemic Lupus International Collaborating Clinics Classification (SLICC) criteria
4. On a stable SLE treatment regimen consisting of any of the following medications for a period of at least 30 days prior to Screening

   * Corticosteroids (<30 mg prednisone or equivalent per day)
   * Hydroxychloroquine or equivalent anti-malarial
   * Other immunosuppressive or immunomodulatory agents including methotrexate, azathioprine, leflunomide, mycophenolate (including mycophenolate mofetil or sodium), cyclophosphasmide, belimumab, calcineurin inhibitors (e.g. tacrolimus, cyclosporine)
5. Willing to perform and comply with all study procedures, including attending clinic visits at Baseline, Month 1, and Month 2 as scheduled

Exclusion Criteria:

1. Rapidly progressive neurologic disease
2. Cognitive dysfunction that might interfere with the capacity to use the ePRO device
3. Any condition that might in the investigator's opinion might preclude completion of the study
4. Current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 1 year prior to Screening
5. Clinical evidence of significant unstable or uncontrolled acute or chronic diseases not caused by SLE (e.g., diabetes, cardiovascular, pulmonary, hematologic, gastrointestinal, neurological, or infectious) which, in the opinion of the Investigator, could confound the results of the study or put the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SLE.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
ePRO Validation | 7 months
  To evaluate measurement equivalence between the two PRO data collection modes - original paper mode versus the ePRO application on a handheld mobile phone for the following PRO's: SF-36 HRQoL questionnaire, the FACIT-F fatigue instrument, and the PtGA. The three PROs will be administered on clinic days by both modes: paper and ePRO. Concurrent results will be compared, and percentage similarities calculated.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (5):
  - Emory University, Atlanta, Georgia
  - Brigham and Women's HospitL, Boston, Massachusetts
  - Northwell Health, Great Neck, New York
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - McMaster University Medical Centre, Hamilton, Ontario
  - University of Western Ontario/St. Joseph's Healthcare, London, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No